CLINICAL TRIAL: NCT00898807
Title: A Multi-Center Randomized Placebo-Controlled Clinical Trial Study of Citalopram for the Treatment of Agitation in Alzheimer's Disease
Brief Title: Citalopram for Agitation in Alzheimer's Disease
Acronym: CitAD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: JHSPH Center for Clinical Trials (Other)
Collaborators: National Institute on Aging (NIA) (NIH); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Dave Shade, Director of CitAD Coordinating Center, Johns Hopkins University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IA0155; R01AG031348 (NIH)
Record Dates: First submitted 2009-05-11; First posted 2009-05-12 (Estimated); Results first posted 2014-06-27 (Estimated); Last update posted 2014-06-27 (Estimated); Status verified 2014-06

CONDITIONS: Alzheimer's Disease; Agitation
Keywords: neuropsychiatric symptoms; aggression; mood lability
MeSH Terms: conditions — Alzheimer Disease; Psychomotor Agitation; Aggression | interventions — Citalopram

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Citalopram and psychosocial intervention (Experimental): Target dose of 30 mg per day of citalopram, oral, and psychosocial intervention
  Interventions: Drug: citalopram
- Placebo and psychosocial intervention (Placebo Comparator): Matching placebo, oral, and psychosocial intervention
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: citalopram — target dose 30mg daily for 9 weeks
  Other Names: Celexa
  Arms: Citalopram and psychosocial intervention
Drug: placebo — daily for 9 weeks
  Arms: Placebo and psychosocial intervention

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of citalopram for agitation in Alzheimer's dementia.

DETAILED DESCRIPTION:
This study is designed to examine the efficacy and safety of citalopram as treatment for clinically significant agitation in Alzheimer's dementia (AD) patients. It will also investigate pharmacogenomic, genetic, and clinical predictors of response to citalopram therapy. The management of agitation is a major priority in treating patients with AD. Non-pharmacologic options have limited effectiveness. Several pharmacologic options have been explored, but findings for anticonvulsants, antipsychotics, and cholinesterase inhibitors are disappointing or associated with questionable risk-benefit ratio. Better pharmacologic options are needed. Selective serotonin reuptake inhibitors (SSRIs) show promise as a treatment for agitation in AD, based on evidence of a link between agitation and brain serotonin system abnormalities in AD patients, and on preliminary clinical data from a single-site, randomized controlled trial (RCT) in which citalopram was superior to perphenazine and placebo.

ELIGIBILITY:
Inclusion criteria

* Probable Alzheimer's disease (National Institute of Neurological and Communicative Disorders and Stroke and the Alzheimer's Disease and Related Disorders Association criteria), with Mini-Mental score of 5-28 inclusive
* A medication for agitation is appropriate, in the opinion of the study physician
* Clinically significant agitation for which either

  1. the frequency of agitation as assessed by the Neuropsychiatric Inventory (NPI) is 'Very frequently', or
  2. the frequency of agitation as assessed by the NPI is 'Frequently' AND the severity of the agitation as assessed by the NPI is 'Moderate', or 'Marked'
* Provision of informed consent for participation in the study by patient or surrogate (if necessary) and caregiver
* Availability of primary caregiver, who spends several hours a week with the patient and supervises his/her care, to accompany the patient to study visits and to participate in the study
* No change to Alzheimer's disease (AD) medications within the month preceding randomization, including starting, stopping, or dosage modifications

Exclusion criteria

* Meets criteria for Major Depressive Episode by Diagnostic and Statistical Manual of Mental Disorders, 4th edition, text revision (DSM-IV (TR)) criteria
* Presence of a brain disease that might otherwise explain the presence of dementia, such as extensive brain vascular disease, Parkinson's disease, dementia with Lewy bodies, traumatic brain injury, or multiple sclerosis
* Psychosis (delusions or hallucinations) requiring antipsychotic treatment in the opinion of the study physician
* Prolonged measure of the time between the start of the Q wave and the end of the T wave in the heart's electrical cycle (QT interval)
* Treatment with citalopram is contraindicated in the opinion of the study physician
* Failure of past treatment with citalopram for agitation after adequate trial at a minimally accepted dose (greater than or equal to 20 mg/day)
* Treatment with a medication that would prohibit the safe concurrent use of citalopram, such as Monoamine oxidases (MAO) inhibitors
* Need for psychiatric hospitalization or suicidal
* Current participation in a clinical trial or in any study that may add a significant burden or affect neuropsychological or other study outcomes
* Current treatment with antipsychotics, anticonvulsants (other than dilantin), other antidepressants (other than trazodone, less than or equal to 50 mg per day at bedtime), benzodiazepines (other than lorazepam), or psychostimulants
* Any condition that, in the opinion of the study physician, makes it medically inappropriate or risky for the patient to enroll in the trial

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 186 (Actual)
Dates: Start 2009-07; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Constantine Lyketsos, MD, MHS, Study Chair — Johns Hopkins University; Lon Schneider, MD, Principal Investigator — University of Southern California Keck School of Medicine Memory and Aging Center; Bruce Pollock, MD, Principal Investigator — Centre for Addiction and Mental Health; Jacobo Mintzer, MD, Principal Investigator — Medical University of South Carolina Alzheimer's Research and Clinical Programs; David Shade, Esq, Principal Investigator — Johns Hopkins University; Davengere Devanand, MD, Principal Investigator — Columbia University; Paul Rosenberg, MD, Principal Investigator — Johns Hopkins University; Daniel Weintraub, MD, Principal Investigator — University of Pennsylvania; Anton Porsteinsson, MD, Principal Investigator — University of Rochester; Jerome Yesavage, MD, Principal Investigator — Stanford University
Locations (8):
- United States (7):
  - University of Southern California Keck School of Medicine Memory and Aging Center, Los Angeles, California
  - VA Palo Alto Health Care System, Palo Alto, California
  - Johns Hopkins University, Baltimore, Maryland
  - Columbia University, New York, New York
  - Monroe Community Hospital, Rochester, New York
  - University of Pennsylvania, Section of Geriatric Psychiatry, Ralston House, Philadelphia, Pennsylvania
  - Medical University of South Carolina Alzheimer's Research and Clinical Programs, Charleston, South Carolina
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

REFERENCES:
- [Background] Drye LT, Ismail Z, Porsteinsson AP, Rosenberg PB, Weintraub D, Marano C, Pelton G, Frangakis C, Rabins PV, Munro CA, Meinert CL, Devanand DP, Yesavage J, Mintzer JE, Schneider LS, Pollock BG, Lyketsos CG; CitAD Research Group. Citalopram for agitation in Alzheimer's disease: design and methods. Alzheimers Dement. 2012;8(2):121-30. doi: 10.1016/j.jalz.2011.01.007. Epub 2012 Feb 1. PMID 22301195
- [Result] Porsteinsson AP, Drye LT, Pollock BG, Devanand DP, Frangakis C, Ismail Z, Marano C, Meinert CL, Mintzer JE, Munro CA, Pelton G, Rabins PV, Rosenberg PB, Schneider LS, Shade DM, Weintraub D, Yesavage J, Lyketsos CG; CitAD Research Group. Effect of citalopram on agitation in Alzheimer disease: the CitAD randomized clinical trial. JAMA. 2014 Feb 19;311(7):682-91. doi: 10.1001/jama.2014.93. PMID 24549548
- [Derived] Drye LT, Spragg D, Devanand DP, Frangakis C, Marano C, Meinert CL, Mintzer JE, Munro CA, Pelton G, Pollock BG, Porsteinsson AP, Rabins PV, Rosenberg PB, Schneider LS, Shade DM, Weintraub D, Yesavage J, Lyketsos CG; CitAD Research Group. Changes in QTc interval in the citalopram for agitation in Alzheimer's disease (CitAD) randomized trial. PLoS One. 2014 Jun 10;9(6):e98426. doi: 10.1371/journal.pone.0098426. eCollection 2014. PMID 24914549

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment activities included chart review, telephone interviews and screens, discussion with physicians, and recruitment in the clinic waiting areas and assisted living facilities affiliated with the clinics. The recruitment period lasted from August 2009 to December 2012.
Groups:
- Citalopram and Psychosocial Intervention: Target dose of 30 mg per day of citalopram, oral, and psychosocial intervention
  citalopram : target dose 30mg daily for 9 weeks
- Placebo and Psychosocial Intervention: Matching placebo, oral, and psychosocial intervention
  placebo : daily for 9 weeks
Period: Overall Study
Arm/Group | Citalopram and Psychosocial Intervention | Placebo and Psychosocial Intervention
Started | 94 | 92
Completed | 86 | 83
Not Completed | 8 | 9
Not completed — Withdrawal by Subject | 5 | 3
Not completed — Family pressure to discontinue | 2 | 2
Not completed — Lost to Follow-up | 1 | 3
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Citalopram and Psychosocial Intervention | Placebo and Psychosocial Intervention | Total
Number analyzed (Participants) | 94 | 92 | 186
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 7 | 13
  >=65 years | 88 | 85 | 173
Age, Continuous [Mean (Standard Deviation); unit: years] | 78 (9) | 79 (8) | 78 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 41 | 85
  Male | 50 | 51 | 101
Region of Enrollment [Number; unit: participants]
  United States | 82 | 79 | 161
  Canada | 12 | 13 | 25

OUTCOME MEASURES:

1. Primary Outcome: NeuroBehavior Rating Scale-- Agitation
Description: NeuroBehavioral Rating Scale- Agitation(NBRS-A) assesses multiple types of psychopathology common in dementia and is based on a seven point Likert scale of increasing severity for each item(i.e., 0=not present, 1=very mild, 2-mild, 3=moderate, 4=moderately severe, 5=severe, 6=extremely severe). The NBRS agitation subscore includes NBRS 'inhibition', 'agitation', and 'hostility'. The range is 0 to 18 points. Higher scores indicate more symptoms.
Time Frame: 9 weeks
Population: The primary analysis was an intention-to-treat analysis; analysis was conducted "as randomized". Data from the 186 randomized participants were used in the analytic model. 167 of the 186 patients had week 9 data on the NBRS.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Citalopram and Psychosocial Intervention | Placebo and Psychosocial Intervention
Number analyzed (Participants) | 90 | 85
units on a scale | 4.33 (0.31) | 5.26 (0.31)
Statistical Analysis 1: Comparison: Citalopram and Psychosocial Intervention vs Placebo and Psychosocial Intervention; Primary assessment of efficacy was based on intention-to-treat comparison of the difference in the NBRS-A scores at week 9 and comparison at week 9 for the CGIC. For the NBRS-A, the study was designed to have 85% power to detect a standardized difference at week 9 of 40% for citalopram compared to placebo at week 9; Test type: Superiority or Other; p = 0.036, Mixed Models Analysis — P-value was not adjusted for multiple comparisons. All p-values are two-sided and p<0.05 was the threshold for statistical significance; Mixed effects model w/ random intercept for patient, visit indicator, treatment by visit interactions and adjusted for baseline NBRS-A & cognition; Mean Difference (Net) = -0.93, 95% CI 2-sided [-1.80 to -0.06] — Negative numbers favor citalopram group

2. Primary Outcome: Modified Alzheimer's Disease Cooperative Study- Clinical Global Impression of Change in Agitation(CGIC)
Description: Modified Alzheimer's Disease Cooperative Study- Clinical Global Impression of Change in agitation(CGIC) accesses clinically significant change in agitation. A trained clinician, blind to treatment assignment, uses a 7-point Likert scale to rate change of each patient along a continuum from "marked improvement"(1), "no change"(4), and "marked worsening"(7). A number of aspects of the agitation is considered such as emotional agitation, mood liability/distress, psychomotor agitation, verbal aggression, and physical aggression. Range is 1-7.
Time Frame: Baseline to 9 weeks
Population: The primary analysis was an intention-to-treat analysis; analysis was conducted "as randomized". Data from the 186 randomized participants were used in the analytic model. 167 of the 186 patients had week 9 data on CGIC.
Measure: Number; unit: percentage moderate/marked improvement
Arm/Group | Citalopram and Psychosocial Intervention | Placebo and Psychosocial Intervention
Number analyzed (Participants) | 86 | 81
percentage moderate/marked improvement | 40 | 26
Statistical Analysis 1: Comparison: Citalopram and Psychosocial Intervention vs Placebo and Psychosocial Intervention; Primary assessment of efficacy was based on intention-to-treat comparison of the difference in the NBRS-A scores at week 9 and comparison at week 9 for the CGIC. For the CGIC proportional odds analysis, the study was designed to have power greater than 80% to detect a difference of 20% between citalopram and placebo in the proportions of patients who improve (or worsen); Test type: Superiority or Other; p = 0.007, Proportional odds — All p-values are two-sided and p <0.05 was the threshold for statistical significance. No adjustments were made for multiple comparisons; estimated treatment effect from the proportional odds model; Odds Ratio (OR) = 2.13, 95% CI 2-sided [1.23 to 3.69] — Positive numbers favors citalopram

3. Secondary Outcome: Cohen-Mansfield Agitation Inventory (CMAI)
Description: CMAI examines several agitated behaviors including verbal, physical agitation, and other behaviors. Sub-items are summed. Range is 14-70. Higher scores indicate more severe symptoms.
Time Frame: 9 weeks
Population: The primary analysis was an intention-to-treat analysis; analysis was conducted "as randomized". Data from the 186 randomized participants were used in the analytic model. 169 of the 186 patients had week 9 data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Citalopram and Psychosocial Intervention | Placebo and Psychosocial Intervention
Number analyzed (Participants) | 90 | 85
units on a scale | 27.7 (6.7) | 28.7 (6.7)

4. Secondary Outcome: Neuropsychiatric Inventory (NPI)-- Agitation Subscore
Description: NPI agitation score is based on responses from an informed caregiver involved in the patient's life. Symptom severity (1=mild, 2=moderate, 3=severe) is multiplied by frequency (1=occasionally, less than once/week; 4 = very frequently, once or more/day or continuously) to obtain the NPI agitation score.Range is 0-12. Higher scores indicate more severe symptoms.
Time Frame: 9 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Citalopram and Psychosocial Intervention | Placebo and Psychosocial Intervention
Number analyzed (Participants) | 90 | 85
units on a scale | 7.8 (2.2) | 8.0 (2.4)

ADVERSE EVENTS:
Description: Adverse events (AEs) are collected systematically on the follow-up visit form; therefore, numbers of participants at risk for AEs reflect at least on follow-up visit form completed. Serious adverse events are often self-reported and can be collected any time throughout the study.
Arm/Group | Citalopram and Psychosocial Intervention | Placebo and Psychosocial Intervention
Serious Adverse Events (participants affected / at risk) | 8/94 | 7/92
Other Adverse Events (participants affected / at risk) | 90/90 | 86/86
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Citalopram and Psychosocial Intervention (N=94) | Placebo and Psychosocial Intervention (N=92)
Mental status change (Psychiatric disorders) | 1 | 2
Sepsis (Infections and infestations) | 1 | 0
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Increased agitation (Psychiatric disorders) | 1 | 2
Fall (Nervous system disorders) | 1 | 1
Hypotension (Cardiac disorders) | 1 | 0
Chest pain (Cardiac disorders) | 1 | 0
Surgical removal of infected plate in wrist (Infections and infestations) | 1 | 0
Lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Abdominal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Citalopram and Psychosocial Intervention (N=90) | Placebo and Psychosocial Intervention (N=86)
Sweating (Nervous system disorders) | 9 | 12
Tremor (Nervous system disorders) | 23 | 16
Dizziness (Nervous system disorders) | 22 | 19
Gait instability (Nervous system disorders) | 50 | 44
Yawning (Nervous system disorders) | 11 | 17
Falls (Nervous system disorders) | 15 | 10
Headache (Nervous system disorders) | 21 | 18
Visual disturbance (Nervous system disorders) | 12 | 14
Somnolence (Psychiatric disorders) | 47 | 42
Insomnia (Psychiatric disorders) | 28 | 39
Anxiety (Psychiatric disorders) | 65 | 66
Deceased libido (Psychiatric disorders) | 14 | 18
Confusion (Psychiatric disorders) | 69 | 72
Suicidal thoughts (Psychiatric disorders) | 6 | 4
Abdominal pain (Gastrointestinal disorders) | 14 | 19
Anorexia (Gastrointestinal disorders) | 40 | 26
Nausea (Gastrointestinal disorders) | 5 | 6
Diarrhea (Gastrointestinal disorders) | 25 | 12
Dry mouth (Gastrointestinal disorders) | 21 | 24
Indigestion (Gastrointestinal disorders) | 23 | 18
Constipation (Gastrointestinal disorders) | 13 | 22
Vomiting (Gastrointestinal disorders) | 5 | 0
Asthenia (Musculoskeletal and connective tissue disorders) | 29 | 30
Muscle pain (Musculoskeletal and connective tissue disorders) | 29 | 34
Joint pain (Musculoskeletal and connective tissue disorders) | 40 | 48
Ejaculatory dysfunction (Reproductive system and breast disorders) | 6/48 | 3/48
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 17 | 9
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 33 | 30
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 27 | 26
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 22 | 22
Sore throat (Respiratory, thoracic and mediastinal disorders) | 7 | 7
Fatigue (General disorders) | 54 | 53
Fever (Infections and infestations) | 9 | 2
Drug allergy (General disorders) | 4 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No